CLINICAL TRIAL: NCT06758869
Title: Effects of Daily Consumption of Processed Pulse-based Food Products on Physiological Responses Related to Energy Metabolism and Metabolic Health
Brief Title: Pulse Revolution: Enhancing Metabolic Health Through the Power of Processed Chickpeas
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Shanon Casperson, Research Biologist, USDA Grand Forks Human Nutrition Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GFHNRC514
Record Dates: First submitted 2024-12-19; First posted 2025-01-06 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Experimental): Base DGA diet with a standardized non-pulse product snack
  Interventions: Other: Control
- Whole Chickpeas (Experimental): Adjusted DGA diet with standardized whole chickpea snack
  Interventions: Other: Whole Chickpeas
- Puréed Chickpeas (Experimental): Adjusted DGA diet with standardized puréed chickpea snack
  Interventions: Other: Puréed Chickpeas
- 100% Chickpea Flour Product (Experimental): Adjusted DGA diet with standardized 100% chickpea flour product snack
  Interventions: Other: 100% Chickpea Flour Product

INTERVENTIONS:
Other: Control — Participants will consume the Base DGA diet with a standardized non-pulse product snack.
  Arms: Control
Other: Whole Chickpeas — Participants will consume an adjusted DGA diet with a standardized whole chickpea snack.
  Arms: Whole Chickpeas
Other: Puréed Chickpeas — Participants will consume an adjusted DGA diet with a standardized puréed chickpea snack.
  Arms: Puréed Chickpeas
Other: 100% Chickpea Flour Product — Participants will consume an adjusted DGA diet with a standardized 100% chickpea flour product snack.
  Arms: 100% Chickpea Flour Product

SUMMARY:
The purpose of this research is to test how processing can affect how one's body uses the nutrients in that food. For this study the researchers are examining how making different food products out of chickpeas, such as hummus or pasta, changes how one's body uses those foods for energy.

DETAILED DESCRIPTION:
The overall objective is to determine the impact of daily consumption of processed pulse-based food products on metabolic health, specifically the physiological responses related to energy metabolism. The primary hypothesis is that consuming a serving of pulses daily for 12 weeks will improve metabolic responses related to energy metabolism, particularly fat oxidation and molecular adaptations related to fat and glucose metabolism, compared to current Dietary Guidelines for Americans (DGA) recommendations. Furthermore, we hypothesize that the degree of processing will influence these metabolic adaptations such that the daily consumption of 100% pulse flour food products will result in the greatest effect on fat oxidation and molecular adaptations related to fat and glucose metabolism followed by the pulse purée which will have a greater effect than the whole cooked pulse (100% pulse flour > purée > whole).

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy adults
* BMI >18.5 or <35 kg/m2 (healthy body weight - class I obesity)
* ability to understand and sign the consent form
* availability of transportation (i.e., participants must provide their own transportation to the Center)
* non-smoking or do not use other tobacco products, including e-cigarettes
* not taking steroid-based medications
* not planning to or currently attempting to gain or lose weight
* not allergic to study foods
* willing to comply with study demands

Exclusion Criteria:

* usual pulse consumption greater than DGA recommendation
* inability or unwillingness to consume any of the provided foods
* more than a 10% change in body weight within the past 2 months
* actively trying to lose weight
* pregnancy or actively trying to get pregnant
* lactation
* uncontrolled hypertension (systolic >160 mmHg or diastolic >100 mmHg)
* diagnosed cardiovascular, pulmonary, skeletal and metabolic diseases
* HbA1c ≥ 5.7%
* complete blood count (CBC) outside of the normal range for a healthy adult
* history of gastrointestinal (GI) disorders (including Celiac's or Crohn's disease, irritable bowel syndrome, acid reflux, ulcerative colitis, chronic constipation or diarrhea, and lactose intolerance)
* using medications known to affect appetite, blood lipids, body composition, body weight, or food intake (appetite control drugs, steroids)
* cannot read or understand English

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Differences in substrate oxidation in response to eating differentially processed pulse-based food products | 12 weels
  Using whole-room calorimetry, measure differences in fat, carbohydrate, and protein oxidation in response to daily consumption of whole chickpeas, pureed chickpeas, or chickpea-flour pasta compared to a control diet.
Change from Baseline in substrate oxidation after consuming differentially processed pulse-based food products for 12 weeks | 12 weeks
  Measure changes in fat, carbohydrate, and protein oxidation in response to consuming whole chickpeas, pureed chickpeas, or chickpea-flour pasta using whole room calorimetry
Determine participant consumption practices and attitudes towards pulse consumption using a validated questionnaire | Baseline
  The questionnaire is designed to assess enjoyment (two items), sensory properties (eight items), perceived cooking abilities (ten items), perceived practical aspects (six items), perceived healthiness (two items), upbringing (two items), social influences (four items), and quality issues (six items) of pulse consumption.

SECONDARY OUTCOMES:
Changes in the colonic microbiota in response to consuming differentially processed pulse-based food products | 12 weeks
  Fecal samples will be collected at Baseline and then again at weeks 4, 8, and 12 to identify how the predominant colon bacteria phyla are effected by consuming whole chickpeas, pureed chickpeas, or chickpea-flour pasta for 12 weeks.
Changes in me metabolic gene expression and metabolites in response to consuming differentially processed pulse-based food products. | 12 weeks
  Blood samples will be collected before and after consuming whole chickpeas, pureed chickpeas, or chickpeas-flour pasta for 12 weeks to identify how consuming these foods effect the expression genes involved with fat metabolism. This will be accomplished by combining the different snapshots provided from pre/post intervention metabolomic, transcriptomic, and proteomic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Shanon Casperson, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Grand Forks Human Nutrition Research Center Current Nutrition Studies — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/docs/nutrition-studies/nutrition-studies/